CLINICAL TRIAL: NCT06776328
Title: Co-creation of Tools for Children and Adolescents with Suicidal Thoughts And/or Behaviour
Acronym: Co-crea K&J
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2024-0211; GE0-1GDF2JA (Other: Flemish government)
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Suicide Prevention; Suicidal Ideation; Suicidal Behaviors
Keywords: co-creation; participatory research; children; adolescents; suicide prevention; suicidal ideation; suicidal behaviour; suicide
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Co-creation meetings (Other): All participants will be invited to participate in the co-creation meetings.
  Interventions: Other: Tools

INTERVENTIONS:
Other: Tools — In the co-creation meetings, developed tools will be presented. Participants will be asked to provide feedback and input to tailor these tools to the needs and preferences of children and adolescents with suicidal thoughts/behavior.

SUMMARY:
Evidence shows that there are very few evidence-based tools or interventions specifically targeting suicidality in children and adolescents. It is crucial to address suicidal thoughts in these populations, as research indicates that discussing suicidality does not increase suicidal behavior but may instead reduce the associated risk. Furthermore, the field of suicide prevention increasingly incorporates digital technologies. Studies suggest that digital interventions targeting suicidality in young people show promise in enhancing knowledge, regulating emotions, developing coping skills, and managing suicidal thoughts and behaviors.

As part of this project, we will develop the following practical tools:

* A creative methodology for professionals to engage children and adolescents in talking about their suicidal thoughts.
* A self-help app for suicidal young people and their support networks. The development process will involve co-creation, with input from children and adolescents playing a central role.

A total of 30 children and adolescents aged 10 to 18 years, who have experienced suicidal thoughts in the past, will participate in this project. The co-creation sessions will be conducted in groups of up to 10 participants. Participants can attend a minimum of 1 and a maximum of 10 sessions, each lasting up to 1.5 hours. The sessions will be facilitated by researchers from VLESP and will take place at a location convenient for participants or in Ghent (the primary location of the research team). If preferred by participants, one or more sessions may also be held online.

For participants who do not wish to join a group, individual sessions can be arranged. Each session will be attended by two researchers, with the potential involvement of professionals specializing in tool development. Several potential developers will be invited to submit proposals for creating the tools, and the selection of the developer will be based on these submissions.

During the sessions, participants will review and evaluate various prototypes of the app. However, the prototypes will not be tested for effectiveness by the young participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 10-18 years
* Proficient in Dutch
* Has experienced suicidal thoughts in the past

Exclusion Criteria (as assessed by the care provider):

* Limited cognitive ability
* Currently experiencing an acute suicidal crisis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Co-creation questions | From enrolment to end of co-creation sessions (10 sessions of 1.5 hours max over the course of the study)
  In the co-creation sessions, participants will be asked about:
  * Current app usage
  * Preferences and needs regarding an app/creative methodology
  * Accessibility and usability of the tools
  * Privacy and confidentiality
  * Social support and community engagement
  * Sensitivity and language
  * Seeking help and professional support
  * Sustained engagement
  * Feedback on tool prototypes
  * Reflections on how they experienced the session

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, PhD, Principal Investigator — Flemish Centre of Expertise in Suicide Prevention, Department of Head and Skin, UGent
Locations (1):
- Flemish Centre of Expertise in Suicide Prevention, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No